CLINICAL TRIAL: NCT03730077
Title: Integrated Biomarker PET/CT Imaging Trial for Assessing Hypoxia in Soft Tissue Sarcomas Using a Novel PET/CT Tracer
Brief Title: FMISO PET/CT Imaging Trial for Assessing Hypoxia in Soft Tissue Sarcomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Left Institution
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 830018
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — fluoromisonidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 18F-MISO PET/CT Test Retest (Experimental): Up to 5 of the 30 intended subjects will participate in a test-retest group that will undergo a second 18F-FMISO scan. Subjects will undergo biopsy as part of their clinical care. Subjects will be asked to consent to allow archived excess tissue to be accessed for the purposes of this study
  Interventions: Drug: 18F-FMISO
- 18F-MISO PET/CT (Experimental): The investigators anticipate enrolling up to 30 subjects who will undergo 18F-FMISO PET/CT.Subjects will undergo biopsy as part of their clinical care. Subjects will be asked to consent to allow archived excess tissue to be accessed for the purposes of this study
  Interventions: Drug: 18F-FMISO

INTERVENTIONS:
Drug: 18F-FMISO — 18F-FMISO PET/CT

SUMMARY:
Subjects with known or suspected primary soft tissue sarcoma of the extremities may be eligible for this study. Subjects may participate in this study if they are at least 18 years of age. Most participants will be receiving care at the clinical practices of the University of Pennsylvania Health System.

Positron emission tomography (PET/CT) imaging will be used to evaluate soft tissue sarcoma hypoxia using an investigational radiotracer, 18F-FMISO Subjects will also undergo an 18F-FDG PET/CT scan close to the time of their initial hypoxia PET/CT to compare in vivo measures of hypoxia to 18F-FDG uptake. The FDG PET/CT may be performed as part of standard clinical care or as a research scan. Both PET/CT scans will occur prior to starting new therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Known or suspected soft tissue sarcoma seen on at least one type of standard imaging (e.g. CT, ultrasound, MRI, or 18F-FDG PET/CT)
2. At least 18 years of age
3. Subjects with local disease or advanced/metastatic disease will be eligible
4. Willing to consent to use of tissue from biopsy or surgery for the purposes of this study
5. Participants must be informed of the investigational nature of this study and be willing and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant at the time of screening will not be eligible for this study; a urine pregnancy test will be performed at screening in women of child-bearing potential
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Hypoxia in FMISO PET/CT | 2 years
  In vivo measures of hypoxia as measured by PET/CT hypoxia tracer (18F-MISO) uptake with PLOD2 expression levels obtained using qRT-PCR in subjects with STS and to identify hypoxia tracer uptake threshold values for in vivo hypoxia based on PLOD2 expression levels

SECONDARY OUTCOMES:
Marker of STS Hypoxia | 2 years
  hypoxia tracer uptake as a marker of STS hypoxia by assessing how in vivo tracer (18F-MISO) T/M uptake ratios correlate with in vitro markers of hypoxia (including HIF-1α, and CAIX) obtained from immunohistochemistry
Relationship of sarcoma hypoxia to glycolysis | 2 years
  The relationship of sarcoma hypoxia to glycolysis using a PET/CT hypoxia tracer (18F-MISO) tumor-to-muscle (T/M) uptake ratios compared to the maximum standardized uptake values (SUVmax) obtained from 18F-FDG PET/CT
Predictors of in vitro PLOD2 expression levels | 2 years
  Best predictors of in vitro PLOD2 expression levels using a PET/CT hypoxia tracer (18F-MISO) and 18F-F-FDG PET/CT uptake values, including HIF-1α and CAIX, and other hypoxia markers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided